CLINICAL TRIAL: NCT00871689
Title: Haploidentical Donor NK Cell Adoptive Therapy and Double T Cell Depleted Umbilical Cord Blood Transplantation With Post-Transplant IL-2 Immune Therapy For Refractory Acute Myeloid Leukemia
Brief Title: Chemotherapy, Total-Body Irradiation, Donor Natural Killer Cell Infusion, Aldesleukin, and UCB Transplant in Treating Patients With Relapsed or Refractory AML
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to graft failure.
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008LS110; MT2008-36 (Other: Blood and Marrow Transplantation Program); 0810M51781 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Results first posted 2012-07-16 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent childhood acute myeloid leukemia; secondary acute myeloid leukemia; childhood acute myeloid leukemia with 11q23 (MLL) abnormalities; childhood acute myeloid leukemia with inv(16)(p13;q22); childhood acute myeloid leukemia with t(15;17)(q22;q12); childhood acute myeloid leukemia with t(16;16)(p13;q22); childhood acute myeloid leukemia with t(8;21)(q22;q22)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Congenital Abnormalities | interventions — aldesleukin; Interleukin-2; Cyclophosphamide; fludarabine phosphate; fludarabine; Cord Blood Stem Cell Transplantation; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- UCBT With Post-Transplant IL-2 (Experimental): Patients receive cyclophosphamide, fludarabine phosphate, total-body irradiation, T cell depleted umbilical cord blood transplantation (UCBT), followed by interleukin-2 (IL-2, aldesleukin) every other day beginning day +3 for a total of 6 doses and again on day +60 every other day for 6 doses.
  Interventions: Biological: aldesleukin; Drug: cyclophosphamide; Drug: fludarabine phosphate; Procedure: umbilical cord blood transplantation; Radiation: total-body irradiation

INTERVENTIONS:
Biological: aldesleukin — IL-2 will be administered (9 million units; 5 million units if weight is less than 45 kg) every other day beginning on day +3 for a total of 6 doses and again on day +60 every other day for 6 doses.
  Other Names: IL-2; interleukin-2
Drug: cyclophosphamide — 60 mg/kg over 1 hour intravenously (IV) on days -7 and -6.
  Other Names: Cytoxan
Drug: fludarabine phosphate — 25 mg/m^2 intravenously (IV) over 1 hour on days -7 through -5.
  Other Names: Fludarabine; Fludara
Procedure: umbilical cord blood transplantation — On day 0, transplantation will occur with double T-cell depleted (TCD) umbilical cord blood (UCB) units
  Other Names: UCBT
Radiation: total-body irradiation — administered on days -5 through -2; 330 cGy daily
  Other Names: TBI

SUMMARY:
RATIONALE: Giving chemotherapy and total-body irradiation before a donor umbilical cord blood stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells and natural killer cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Giving interleukin-2 (IL-2, aldesleukin) after transplant may stimulate the natural killer cells to kill any remaining cancer cells.

PURPOSE: This phase II trial is studying the side effects of giving combination chemotherapy together with total-body irradiation followed by interleukin-2 (IL-2, aldesleukin), and umbilical cord blood transplant and to see how well it works in treating patients with relapsed or refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the rate of neutrophil engraftment and grade III-IV acute graft-versus-host disease (GVHD) following a T cell depleted (TCD) umbilical cord blood (UCB) transplantation without post-transplant immunosuppression followed by administration of interleukin-2 (IL-2, aldesleukin) (every other day) days +3 to +13 to expand NK cells in vivo.

Secondary

* To evaluate the safety of this regimen as assessed by monitoring the rates of graft failure, acute GVHD, and transplant-related mortality (TRM).
* To perform quantitative, phenotypic, and functional assessments of the in vivo expanded UCB-derived NK cells on (day +72).
* To assess clinical disease response (leukemia clearance and complete remission) and survival duration in these patients.
* To evaluate the tolerability of aldesleukin in these patients.
* To evaluate the tolerance of IL-2

OUTLINE:

* Preparative regimen: Patients receive fludarabine phosphate intravenously (IV) over 1 hour on days -7 to -5 and cyclophosphamide IV on days -7 and -6. Patients undergo total-body irradiation twice daily on days -5 to -2.
* Transplantation: Patients undergo T-cell depleted umbilical cord blood (UCB) transplantation on day 0.
* IL-2 (Aldesleukin) therapy: Patients receive aldesleukin subcutaneously on days +3 6 doses every other day) and +60 (6 doses every other day).

Patients are followed periodically for up to 2 years after transplant.

ELIGIBILITY:
Inclusion Criteria:

* Aged 0 to 45 years who meet one of the following criteria:

  * Primary induction failure defined as no complete remission (CR) after two or three induction cycles (no blast limit).
  * Relapsed acute myeloid leukemia (AML) with low disease burden

    * For patients 19 through 45 years of age: must have less than 10% marrow blasts at time of enrollment for patients who did not receive re-induction or measured at least 28 days from the start of re-induction therapy. Patients who have relapsed more than 12 months following a prior hematopoietic cell transplant (HCT) and did not reach CR following one re-induction cycle but have less than 10% marrow blasts are eligible.
    * For patients 0 through 18 years of age: must have less than 50% marrow blasts after no more than 3 induction attempts
  * CR3 or greater. This will include CRp defined as CR without platelet recovery to 100,000/mcL.
  * CR1 or CR2 with high risk features (therapy induced, prior myelodysplastic syndrome (MDS) or myeloproliferative disease (MPD), high risk cytogenetic or molecular phenotype) with no available alternate (sibling, URD or UCB) donors.
* Patients with prior central nervous system (CNS) involvement are eligible provided that it has been treated and is in remission. CNS therapy (chemotherapy or radiation) should continue as medically indicated during the protocol.
* Have acceptable organ function within 14 days of enrollment defined as:

  * Renal: creatinine ≤ 2.0 mg/dL (adult patients) or calculated creatinine clearance > 40 ml/min (pediatric patients)
  * Hepatic: bilirubin, AST/ALT, ALP ≤ 5 x upper limit of normal
  * Pulmonary function: DLCOcorr > 50% of normal, (oxygen saturation [>92%] can be used in child where PFT's cannot be obtained)
  * Cardiac: left ventricular ejection fraction ≥ 45%
* Karnofsky score (adults) > 70% or Lansky score > 50% (pediatrics)
* Women of childbearing potential must agree to use adequate contraception (diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.) for the duration of treatment.
* All patients will be questioned about prior exposure to antibody therapy (including OKT3, rituximab, trastuzumab, and gemtuzumab) without affect to eligibility. Patients with prior exposure will have a blood sample collected for human anti-mouse antibody (HAMA). For patients with no prior antibody therapy exposure, no further action will be taken.
* Not receiving prednisone or other immunosuppressive medications
* Voluntary written consent

Exclusion Criteria:

* Active infection at time of enrollment or documented fungal infection within 3 months
* Evidence of HIV infection or known HIV positive serology
* Pregnant or breast feeding. The agents used in this study may be teratogenic to a fetus and there is no information on the excretion of agents into breast milk. All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy.
* If ≤ 18 years old, prior myeloablative transplant within the last 6 months. If > 18 years old prior myeloablative allotransplant or autologous transplant
* Extensive prior therapy including > 12 months of any alkylator chemotherapy (etoposide >100 mg/m^2 x 5 days, cyclophosphamide >1 gm/m^2 or mitoxantrone >8 gm/m^2) delivered at 3-4 week intervals or > 6 months alkylator therapy (as above) with extensive radiation (determined by Radiation Oncology, e.g. mantle irradiation for Hodgkin's) and/or prior radiation therapy that makes a patient ineligible for total body irradiation (TBI).

Criteria for Second Course of IL-2 (begin day +60):

* No Graft-Versus-Host Disease (GVHD), active infection or any other severe medical co-morbidity
* Absolute neutrophil count (ANC) > 1000 without growth factor support
* No grade 4 toxicity (except fevers) attributed to IL-2 during course #1

Max Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2009-01; Primary Completion 2010-03 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. Verneris, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Children's Hospital - Fairview, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study entry was open to patients aged 0 to 45 years regardless of gender or ethnic background at the University of Minnesota, Masonic Cancer Center.
Groups:
- Patients Receiving Double Umbilical Cord Blood Transplant: Patients that receive myeloablative preparative regimen (allopurinol 300 mg by mouth Day -8 through +14; fludarabine 25 mg/m^2 intravenously on days -7 through -5; cyclophosphamide 60 mg/kg intravenously on days -7 and -6; total body irradiation 165 cGy*2 on days -4 through -2), 2 units T cell depleted umbilical cord blood transplant on day 0, followed by IL-2 every other day beginning day +3 and day +60 for a total of 6 doses.
Period: Overall Study
Arm/Group | Patients Receiving Double Umbilical Cord Blood Transplant
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Receiving Double Umbilical Cord Blood Transplant
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.5 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Neutrophil Engraftment
Description: Number of patient with absolute neutrophils >500*10^8/kg by 42 days post transplant.
Time Frame: Day 42
Measure: Number; unit: Participants
Arm/Group | Patients Receiving Double Umbilical Cord Blood Transplant
Number analyzed (Participants) | 2
Participants | 1

2. Secondary Outcome: Incidence of Primary Graft Failure
Description: Incidence of graft failure defined as an absolute neutrophil count of less than 500/uL and a bone marrow that is less than 5% cellular (marrow aplasia) on day 42.
Time Frame: Day 42
Measure: Number; unit: Participants
Arm/Group | Patients Receiving Double Umbilical Cord Blood Transplant
Number analyzed (Participants) | 2
Participants | 1

3. Secondary Outcome: Number of Patients With Acute Graft-Versus-Host (GVHD) Disease
Description: Number of patients with any grade of GVHD. Graft-versus-host disease (GVHD) is a complication that can occur after a stem cell or bone marrow transplant in which the newly transplanted material attacks the transplant recipient's body.
  Acute GVHD usually happens within the first 3 months after transplant.
Time Frame: Day 100 Post Transplant
Measure: Number; unit: participants
Arm/Group | Patients Receiving Double Umbilical Cord Blood Transplant
Number analyzed (Participants) | 2
participants | 1

4. Secondary Outcome: Number of Patients With Transplant-Related Death (TRD)
Description: Number of patients whose death is related to study treatment received. TRD is defined as the number of patients that die without prior relapse.
Time Frame: 1 Year Post Transplant
Measure: Number; unit: Participants
Arm/Group | Patients Receiving Double Umbilical Cord Blood Transplant
Number analyzed (Participants) | 2
Participants | 1

5. Secondary Outcome: Number of Patients With Complete Remission of Disease
Description: Disease response will be measured by rate of leukemic clearance (clearance of blasts in blood at timepoint 0) and complete remission (less than 5% blasts and recovery of hematopoiesis).
Time Frame: Day 100
Measure: Number; unit: Participants
Arm/Group | Patients Receiving Double Umbilical Cord Blood Transplant
Number analyzed (Participants) | 2
Participants | 1

6. Primary Outcome: Number of Patients With Grade III-IV Acute Graft-Versus-Host (GVHD) Disease
Description: Number of patients with Grade III-IV GVHD. Graft-versus-host disease (GVHD) is a complication that can occur after a stem cell or bone marrow transplant in which the newly transplanted material attacks the transplant recipient's body.
  Acute GVHD usually happens within the first 3 months after transplant.
Time Frame: Day 100 Post Transplant
Measure: Number; unit: participants
Arm/Group | Patients Receiving Double Umbilical Cord Blood Transplant
Number analyzed (Participants) | 2
participants | 0

7. Secondary Outcome: Median Overall Survival
Description: Average number of days the patients were alive after receiving UCB transplantation.
Time Frame: Month 6
Measure: Median (Full Range); unit: Days
Arm/Group | Patients Receiving Double Umbilical Cord Blood Transplant
Number analyzed (Participants) | 2
Days | 98.5 [98 to 99]

8. Secondary Outcome: Number of Patients With Successful Natural Killer Expansion
Description: Successful in vivo donor NK cell expansion will be defined as an absolute circulating donor-derived NK cell count of >100 cells/μl.
Time Frame: Day 72 Post Transplant
Measure: Number; unit: participants
Arm/Group | Patients Receiving Double Umbilical Cord Blood Transplant
Number analyzed (Participants) | 2
participants | 1

ADVERSE EVENTS:
Time Frame: Patients were followed from Day 1 up to death ( within 6 months).
Arm/Group | Patients Receiving Double Umbilical Cord Blood Transplant
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Receiving Double Umbilical Cord Blood Transplant (N=2)
Death (General disorders) | 2 (2)
Leukoencephalopathy (Blood and lymphatic system disorders) | 1 (2)
CNS Demyelinating Disease (Nervous system disorders) | 1 (2)
Progressive Disease (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Receiving Double Umbilical Cord Blood Transplant (N=2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever (General disorders) | 2 (7)
Chills (Nervous system disorders) | 2 (6)
Hypertension (Cardiac disorders) | 1 (3)
Hypotension (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 2 (6)
Edema (Endocrine disorders) | 2 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Injection site reaction (Skin and subcutaneous tissue disorders) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (3)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (2)
Sweats (Nervous system disorders) | 1 (3)
Vomiting (Gastrointestinal disorders) | 1 (2)

LIMITATIONS AND CAVEATS:
Quantitative, phenotypic and functional assessment of the in vivo expanded UCB-derived NK cells on Day 72 were not performed. Patients were not well enough to provide research samples.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes